CLINICAL TRIAL: NCT04647708
Title: A Phase Ib, Randomized, Double-blind, Placebo Controlled Study to Evaluate the Safety and Pharmacokinetics of Multiple Ascending Doses of M5049 Administered Orally in SLE and CLE Participants Treated With Standard of Care
Brief Title: Study of M5049 in CLE and SLE Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MS200569_0004; 2020-003118-11 (EudraCT Number)
Record Dates: First submitted 2020-11-23; First posted 2020-12-01 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Systemic Lupus Erythematosus; Cutaneous Lupus Erythematosus
Keywords: Lupus Erythematosus, Systemic; Lupus Erythematosus, Cutaneous; Autoimmune Diseases
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Erythematosus, Cutaneous; Autoimmune Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Part A (Cohort 1): M5049 Dose A (Experimental)
  Interventions: Drug: M5049
- Part A (Cohort 2): M5049 Dose B (Experimental)
  Interventions: Drug: M5049
- Part A (Cohort 3): M5049 Dose C (Experimental)
  Interventions: Drug: M5049
- Part A (Cohort 4): M5049 Dose D (Experimental)
  Interventions: Drug: M5049
- Part A: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Part B (Cohort 5): M5049 Dose E (Experimental)
  Interventions: Drug: M5049
- Part B: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: M5049 — Participants will receive low oral dose of M5049, twice daily in Part A.
  Arms: Part A (Cohort 1): M5049 Dose A
Drug: M5049 — Participants will receive ascending oral dose of M5049, twice daily in Part A.
  Arms: Part A (Cohort 2): M5049 Dose B; Part A (Cohort 3): M5049 Dose C; Part A (Cohort 4): M5049 Dose D
Drug: M5049 — Participants will receive high oral dose of M5049, twice daily in Part B.
  Arms: Part B (Cohort 5): M5049 Dose E
Drug: Placebo — Participants will receive placebo matched to M5049.
  Arms: Part A: Placebo; Part B: Placebo

SUMMARY:
This study is to evaluate the safety, tolerability and pharmacokinetics (PK) of orally administered M5049 in participants with systemic lupus erythematosus (SLE) or cutaneous lupus erythematosus (CLE).

ELIGIBILITY:
Inclusion Criteria:

* Active systemic lupus erythematosus (SLE) with a Cutaneous lupus erythematosus disease area and activity index (CLASI-A) greater than or equal to [>= ] 6 and/or at least one active SLE clinical manifestation according to Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K)
* Active cutaneous lupus erythematosus (CLE) (subacute cutaneous lupus erythematosus and/or discoid lupus erythematosus) with a CLASI-A >= 6
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Autoimmune or rheumatic disease other than SLE or CLE
* Dermatological diseases other than cutaneous manifestations of SLE or CLE
* Uncontrolled medical conditions including significant cardiovascular events, active lupus nephritis, and active neurological disorder
* Ongoing or active clinically significant viral, bacterial or fungal infection
* History of uncontrolled seizures or other neurological disorder
* History of or positive for human immunodeficiency virus, hepatitis C virus, or hepatitis B virus
* History of malignancy
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
Part A: Cohort 1 and 2: Number of Participants with Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs and Adverse Event of Special Interest (AESI), TEAEs Leading to Permanent Treatment Discontinuation and Treatment-Related TEAEs | Up to Day 102
Part A: Cohort 3 and 4; Part B: Cohort 5: Number of Participants with Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs and Adverse Event of Special Interest (AESI), TEAEs Leading to Permanent Treatment Discontinuation and Treatment-Related TEAEs | Up to Day 186
Part A: Cohort 1 and 2: Number of Participants with Treatment-Emergent Adverse Events (TEAEs) Based on Severity | Up to Day 102
Part A: Cohort 3 and 4; Part B: Cohort 5: Number of Participants with Treatment-Emergent Adverse Events (TEAEs) Based on Severity | Up to Day 186
Part A: Cohort 1 and 2: Number of Participants with Clinically Significant Changes from Baseline in Laboratory Parameters, Vital Signs, Electroencephalogram (EEG) and Electrocardiogram (ECG) Findings | Up to Day 102
Part A: Cohort 3 and 4; Part B: Cohort 5: Number of Participants with Clinically Significant Changes from Baseline in Laboratory Parameters, Vital Signs, Electroencephalogram (EEG) and Electrocardiogram (ECG) Findings | Up to Day 186
Part A: Cohort 1 and 2: Number of Participants with Confirmed Signs and Symptoms of Prodromal Seizure | Up to Day 102
Part A: Cohort 3 and 4; Part B: Cohort 5: Number of Participants with Confirmed Signs and Symptoms of Prodromal Seizure | Up to Day 186
Part A: Cohort 1 and 2: Number of Participants with Suicidal Behavior and Suicidal Ideation as Assessed by Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to Day 102

SECONDARY OUTCOMES:
Part A and Part B: Maximum Observed Plasma Concentration (Cmax) of M5049 | Pre-dose up to Day 85 for Cohort 1 and 2 of Part A, up to Day 169 for Cohort 3, 4 of Part A and Cohort 5 of Part B
Part A and Part B: Dose Normalized Maximum Observed Plasma Concentration (Cmax/Dose) of M5049 | Day 1 and Day 29
Part A and Part B: Time to Reach Maximum Plasma Concentration (tmax) of M5049 | Pre-dose up to Day 85 for Cohort 1 and 2 of Part A, up to Day 169 for Cohort 3, 4 of Part A and Cohort 5 of Part B
Part A and Part B: Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Sampling Time (AUC0-t) of M5049 | Pre-dose up to Day 85 for Cohort 1 and 2 of Part A, up to Day 169 for Cohort 3, 4 of Part A and Cohort 5 of Part B
Part A and Part B: Dose Normalized Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Sampling Time (AUC0-t/Dose) of M5049 | Day 1 and Day 29
Part A and Part B: Accumulation Ratio for Maximum Observed Plasma Concentration (Racc Cmax) of M5049 | Pre-dose up to Day 85 for Cohort 1 and 2 of Part A, up to Day 169 for Cohort 3, 4 of Part A and Cohort 5 of Part B
Part A and Part B: Elimination Rate Constant (Lambda z) of M5049 | Day 1 and Day 29
Part A and Part B: Apparent Terminal Half-life (t1/2) of M5049 | Day 1 and Day 29
Part A and Part B: Area Under the Plasma Concentration-Time Curve From Time Zero to 12 Hours Post-Dose (AUC0-12h) of M5049 | Day 29
Part A and Part B: Dose Normalized Area Under Plasma Concentration-Time Curve from Time Zero to 12 Hours Post-Dose (AUC0-12h/Dose) of M5049 | Day 29
Part A and Part B: Total Body Clearance (CL/f) of M5049 | Day 1
Part A and Part B: Apparent Volume of Distribution (Vz/f) of M5049 | Day 1
Part A and Part B: Area Under Plasma Concentration-Time Curve from Time Zero Extrapolated to Infinity (AUC0-inf) of M5049 | Day 1
Part A and Part B: Dose Normalized Area Under Plasma Concentration-Time Curve from Time Zero Extrapolated to Infinity (AUC0-inf/Dose) of M5049 | Day 1
Part A and Part B: Change from Baseline in Cutaneous Lupus Erythematosus Disease Area and Activity Index (CLASI-A) | Baseline (Day 1) through Day 85 for Cohort 1 and 2 of Part A, Day 169 for Cohort 3, 4 of Part A and Cohort 5 of Part B
Part A and Part B: Change from Baseline in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) | Baseline (Day 1) through Day 85 for Cohort 1 and 2 of Part A, Day 169 for Cohort 3, 4 of Part A and Cohort 5 of Part B
Part A and Part B: Change from Baseline in 28-Joint Count | Baseline (Day 1) through Day 85 for Cohort 1 and 2 of Part A, Day 169 for Cohort 3, 4 of Part A and Cohort 5 of Part B
Part A and Part B: Change from Baseline in Physician Global Assessment (PGA) Score | Baseline (Day 1) through Day 85 for Cohort 1 and 2 of Part A, Day 169 for Cohort 3, 4 of Part A and Cohort 5 of Part B

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (12):
- Bulgaria (4):
  - Medical center Medconsult Pleven OOD, Pleven
  - Medical Center-1-Sevlievo EOOD, Sevlievo
  - Military Medical Academy - MHAT - Sofia, Sofia
  - UMHAT "Sv. Ivan Rilski", EAD, Sofia
- Germany (2):
  - SocraTec R&D GmbH, Erfurt
  - Fraunhofer ITMP (Fraunhofer Institute for Translational Medicine and Pharmacology), Frankfurt
- ARENSIA Exploratory Medicine Phase I Unit, Clinical Republican Hospital, Chisinau, Moldova
- PHI University Clinic of Rheumatology Skopje, Skopje, North Macedonia
- Spain (3):
  - Hospital Universitario Nuestra Señora de Valme, Seville
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario Rio Hortega - Servicio de Medicina Interna, Valladolid
- Medical Center of Limited Liability Company "Harmoniya krasy", Department of clinical trials, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website https://bit.ly/IPD21

REFERENCES:
- [Derived] Witte T, Fernandez-Ruiz R, Abramova N, Weinelt D, Moreau F, Klopp-Schulze L, Shaw J, Denis D, Wenzel J. Enpatoran, a first-in-class, selective, orally administered toll-like receptor 7/8 inhibitor, in systemic and cutaneous lupus erythematosus: results from a randomised, placebo-controlled phase Ib study. Lupus Sci Med. 2025 Oct 23;12(2):e001705. doi: 10.1136/lupus-2025-001705. PMID 41136221
- [Derived] Klopp-Schulze L, Shaw JV, Dong JQ, Khandelwal A, Vazquez-Mateo C, Goteti K. Applying Modeling and Simulations for Rational Dose Selection of Novel Toll-Like Receptor 7/8 Inhibitor Enpatoran for Indications of High Medical Need. Clin Pharmacol Ther. 2022 Aug;112(2):297-306. doi: 10.1002/cpt.2606. Epub 2022 May 21. PMID 35390178
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200569_0004
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html